CLINICAL TRIAL: NCT04442763
Title: Assessment of Dental Implants Stability After Using Osseodensification Method Versus Conventional Drilling in the Posterior Maxilla: A Randomized Clinical Trial
Brief Title: The Effect of Osseodensification on Implant Stability in Posterior Maxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Amr Abdel Raouf, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sara89
Record Dates: First submitted 2020-06-15; First posted 2020-06-23 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Implant Stability
Keywords: Osseodensification; Densah burs; conventional drilling; implant stability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: the statistician will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Densah burs (Experimental): Osseodensification using Densah burs
  Interventions: Device: Densah Burs
- Standard drills (Active Comparator): conventional drilling using standard drills
  Interventions: Device: Standard drills

INTERVENTIONS:
Device: Densah Burs — osseodensification method
  Arms: Densah burs
Device: Standard drills — conventional drilling
  Arms: Standard drills

SUMMARY:
Implants will be placed in posterior maxilla using two drilling methods; the osseodensification technique and conventional drilling protocols. Implant stability will be measured after implant placement , 1,2,3,4,6 and 8 weeks and 3 months later. Insertion torque will be evaluated at the termination of implant placement and crestal bone loss will be measured post-implant insertion, after 3 months and after 6 and 12 months of loading. Post-operative pain and patients' satisfaction will be assessed as well. implant survival will be assessed at the end of the follow up period

ELIGIBILITY:
Inclusion Criteria:

* Age: >18 years; medically free,
* Partially edentulous patients in maxillary posterior area (premolar-molar area)
* Sufficient ridge height
* Sufficient ridge width
* Adequate soft tissue biotype.
* Patients with adequate inter-arch space for placement of implant prosthetic part.
* Cooperative patients with good oral hygiene
* Patients who accept to sign an informed consent.

Exclusion Criteria:

* Active periodontal diseases
* Parafunctional habits.
* History of radiation therapy to the head and neck
* Bone augmentation to implant site
* Smoking
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Implant stability | immediately post-implant insertion, 1,2,3,4,6,8 weeks and 3 months
  Implant stability will be measured using Osstell (Resonance Frequency Analysis). the measurement unit is Implant stability quotient (ISQ) (range 1-100)

SECONDARY OUTCOMES:
Crestal bone loss | immediately post-implant insertion - 3 months- 6 and 12 months post-loading
  Standardized periapical digital radiographs
Insertion torque | at the termination of implant insertion
  torque wrench

CONTACTS AND LOCATIONS:
Overall Officials: Omnia Aboul Dahab, Study Director — Professor, Faculty of Dentistry, Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Abdelraouf SA, Dahab OA, Mostafa B, Kenawy SM, Tawfik OK. Implant stability in the posterior maxilla: clinical and radiographic comparison of osseodensification and conventional drilling: a randomized clinical trial. Clin Oral Investig. 2025 Sep 29;29(10):480. doi: 10.1007/s00784-025-06526-8. PMID 41016918